CLINICAL TRIAL: NCT04688034
Title: Phase I Clinical Trial of CBP/Beta-catenin Inhibitor OP-724 in Liver Cirrhosis Patients Caused by HIV/HCV Co-infection with Hemophilia. (OP-724-H101)
Brief Title: Safety and Tolerability Study of OP-724 in Liver Cirrhosis Patients by HIV/HCV with Hemophilia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kiminori Kimura, MD (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government); Ohara Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Kiminori Kimura, MD, Head, Department of Hepatology, Komagome Hospital
Organization: Komagome Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OP-724-H101; jRCT2031200266 (Other: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2020-12-21; First posted 2020-12-29 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Liver Cirrhosis
Keywords: Liver Cirrhosis; Hemophilia; HIV/HCV co-infection
MeSH Terms: conditions — Liver Cirrhosis; Hemophilia A | interventions — ICG 001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OP-724 400 mg / 20 mL / vial (20 mg / mL) (Experimental): Dose: [Cohort 1] 140 mg/m2/4 hours (starting dose) , [Cohort 2] 280 mg/m2/4 hours
  Administration method: In the single administration, the safety of concomitant use with the investigational drug and antiretroviral drug will be confirmed and then the cycle administration will be started. For the single administration, at 14 days before the first cycle of administration, the dose planned for the first cycle with continuous intravenous administration for 4 hours will be administrated once. When an integrase inhibitor is used in combination as a key drug for antiretroviral drugs, it should be administered at the same time as the start of investigational drug administration only after the single administration. For the cycle administration, the continuous intravenous administration for 4 hours twice a week is defined as one cycle, and 12 cycles (12 weeks in total) will be performed.
  Interventions: Drug: OP-724

INTERVENTIONS:
Drug: OP-724 — Twice a week for 4 hours continuous intravenous administration of OP-724.
  Other Names: CBP-beta-catenin inhibitor; PRI-724 (former name)

SUMMARY:
To evaluate the safety and tolerability of OP-724 in liver cirrhosis patients caused by HIV/HCV co-infection with hemophilia.

DETAILED DESCRIPTION:
This trial is an uncontrolled, open-label, single-center phase I study in liver cirrhosis patients caused by human immunodeficiency virus (HIV)/hepatitis C virus (HCV) co-infection with hemophilia.

Liver cirrhosis patients due to co-infection of HIV and HCV with hemophilia who have a Child-Pugh classification of A or B are included. OP-724 is intravenously administered twice a week (4 hours) for 12 weeks as an administration schedule.

At 14 days before the administration of the first cycle, the dose planned for the first cycle will be administered once by continuous intravenous administration for 4 hours, and the safety and pharmacokinetics will be evaluated from the day of administration to the day after the administration. If an integrase inhibitor is used in combination as a key drug for antiretroviral drugs, its pharmacokinetics will be evaluated at the same time.

A dose escalation study with 2 doses (cohort 1: 140 mg/m2/4hr (starting dose), cohort 2: 280 mg/m2/4hr) will be conducted, and 3 patients in each cohort will be enrolled. Comprehensively investigate the safety and pharmacokinetic data after OP-724 administration, and evaluate the safety and tolerability of OP-724 administration.

ELIGIBILITY:
Inclusion Criteria:

1. Hemophilia patients with liver cirrhosis caused by HIV/HCV co-infection that fall under the following 1) and 2).

1. HIV-RNA positive in serum or HIV antibody positive patients (the amount of HIV-RNA in the blood at the time of screening is less than 200 copies/mL, and the number of CD4 positive T lymphocytes can be maintained at 200/micro L or more).
2. HCV-RNA positive in serum or HCV antibody positive patients (regardless of the amount of viral and treatment).

2. Patients with Child-Pugh class A or B.

3. Patients who meet at least one of 1) to 3) for diagnosis of liver cirrhosis.

1. FIB-4 index value is 3.25 or higher.
2. Liver hardness value by FibroScan is 11.8 kPa or more.
3. Abdominal CT scan shows changes in liver shape and/or portal hypertension symptoms.

4. Patients who meet any of 1) to 3) for anti-HCV therapy.

1. Patients who have not reached the sustained virological response (SVR) * with the direct acting antivirals (DAA) therapy. * SVR shall be as SVR12 (persistent virus negative at 12 weeks after the end of administration).
2. Patients who have difficulty in performing DAA therapy.
3. Patients who have passed 24 weeks or more after achieving SVR* with DAA therapy or IFN therapy.

5. Patients with Performance Status 0-2.

6. Male patients aged 20 to under 75 at the time of obtaining written consent.

7. Patients who provided voluntary written consent to participate in this clinical trial.

Exclusion Criteria:

1. Patients who have cirrhosis due to causes other than HCV, and patients whose cause of cirrhosis is unknown.
2. Patients with esophagogastric varices who are judged to require treatment by endoscopy at the time of screening.
3. Patients with complication or with previous history of primary liver cancer (excluding patients who have been for more than 1 year after hepatoma removing operation or radiofrequency ablation etc.).
4. Patients with complication or with previous history of malignant tumor (within 3 years before screening).However, except for the following diseases: treated basal cell carcinoma, treated lung carcinoma in situ, or well-controlled superficial (non-invasive) bladder cancer.
5. Patients with active AIDS index disease requiring treatment.
6. Patients for whom HBV, HTLV-1 active viral infection or syphilis infection cannot be ruled out.
7. Serum creatinine level: Patients over 1.5 times the upper limit of the facility reference value.
8. Patients with complications with uncontrolled diabetes, hypertension or heart failure.
9. Patients with psychiatric disorders that may affect the conduct of clinical trial.
10. Patients with or have a history of serious allergies to contrast agent.
11. Patients who have not passed the following period at the time of registration and after the end of anti-HCV therapy.

    * IFN preparation 12 weeks after the last administration
    * Ribavirin preparation 16 weeks after the last administration
    * 16 weeks after the last administration of DAA
12. Patients whose dosage and administration have been changed within 12 weeks prior to registration if the following treatments have been given.

    * Liver cirrhosis
    * HIV
13. Patients with a history of drug or alcohol intoxication within 5 years prior to obtaining written consent, or patients with a history of drug or alcohol abuse within the last 1 year.
14. Patients who participated in other clinical trials within 30 days before obtaining written consent and used or had used investigational drugs or investigational medical devices.
15. Patients who have undergone liver transplantation or other organ transplantation (including bone marrow transplantation) and patients who have difficulty in intravenous administration.
16. Male patients who do not consent to contraception from the time of consent acquisition to 12 weeks after the end of study drug administration.
17. In addition, patients who are judged by the investigator or sub-investigator to be ineligible for this study.

Ages: 20 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events (Side Effects) | 28 days after the last administration of OP-724.
  Occurrence rate of serious adverse events whose causal relationship with the investigational drug cannot be ruled out (side effects). The data will be aggregated by each cohort.

SECONDARY OUTCOMES:
Adverse Events | 28 days after the last administration of OP-724.
  Occurrence rate of adverse events. The data will be aggregated by each cohort, seriousness and severity.
Side Effects | 28 days after the last administration of OP-724.
  Occurrence rate of side effects.
Parameters on Pharmacokinetics (OP-724 and C-82): Maximum Plasma Concentration (Cmax) | Single administration part: pre-dose and post-dose at 0.5, 1, 2, 4, 5, 9 and 24 hours.
  Cmax of OP-724 and C-82 will be determined.
Parameters on Pharmacokinetics (OP-724 and C-82): Area Under the Curve from 0 to 24 hours (AUC0-24h) | Single administration part: pre-dose and post-dose at 0.5, 1, 2, 4, 5, 9 and 24 hours.
  AUC0-24 of OP-724 and C-82 will be determined.
Parameters on Pharmacokinetics (OP-724 and C-82): Time to Maximum Plasma Concentration (Tmax) | Single administration part: pre-dose and post-dose at 0.5, 1, 2, 4, 5, 9 and 24 hours.
  Tmax of OP-724 and C-82 will be determined.
Parameters on Pharmacokinetics (OP-724 and C-82): t1/2 | Single administration part: pre-dose and post-dose at 0.5, 1, 2, 4, 5, 9 and 24 hours.
  t1/2 of OP-724 and C-82 will be determined.
Drug Concentration (OP-724 and C-82) in Plasma | A) Single administration part: pre-dose and post-dose at 0.5, 1, 2, 4, 5, 9 and 24 hours. B) Continuous administration part: pre-dose and post-dose at 4 hours on Day 1 and 4 in Cycle 1, 5, 9 and 12 (each cycle is 7days).
  Graphing with time course of drug concentration.
Drug Concentration (Integrase inhibitor) in Plasma | A) Single administration part: pre-dose and post-dose at 2, 4, 9 and 24 hours. B) Continuous administration part: pre-dose on Day 1 in Cycle 5, 9 and 12 (each cycle is 7days).
  Graphing with time course of drug concentration.
Blood HIV-RNA Level | Baseline, Cycle5Day1, Cycle9Day1 and up to 12 weeks after administration (each cycle is 7days).
  Amount of change in blood HIV-RNA level from baseline at each measurement time point.
CD4 Positive T Lymphocyte Count | Baseline, Cycle5Day1, Cycle9Day1 and up to 12 weeks after administration (each cycle is 7days).
  Amount of change in CD4 positive T lymphocyte count from baseline at each measurement time point.
FibroScan | Baseline and 12 weeks after administration
  Amount of change from baseline in the measured value of liver tissue hardness by FibroScan at 12 weeks after administration.
FIB-4 Index | Baseline and 12 weeks after administration
  Amount of change from baseline in FIB-4 index at 12 weeks after administration.
APRI | Baseline and 12 weeks after administration
  Amount of change from baseline in APRI at 12 weeks after administration.
Child-Pugh Score | Baseline and 12 weeks after administration
  Amount of change from baseline in Child-Pugh Score at 12 weeks after administration. Child Pugh score (scale range 5-15 points, the severity increases sequentially from 5 to 15 points) is obtained by adding the score for each parameter (hepatic encephalopathy, ascites, bilirubin, albumin, PT). Based on the total points score (Child-Pugh Score) of each diagnostic parameter shown above, the severity of the disease is classified into Grades A to C shown below.
  * Grade A: 5-6 points -> Compensated cirrhosis
  * Grade B: 7-9 points -> Decompensated cirrhosis
  * Grade C: 10-15 points -> Decompensated cirrhosis
MELD Score | Baseline and 12 weeks after administration
  Amount of change from baseline in MELD score at 12 weeks after administration.
  The Model for End-Stage Liver Disease (MELD) is a scoring system for assessing the severity of chronic liver disease and uses the subject's values for total bilirubin, serum creatinine, and the international normalized ratio (INR) for prothrombin time to predict survival. MELD is calculated according to the following formula:
  * MELD score = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43

CONTACTS AND LOCATIONS:
Overall Officials: Kiminori Kimura, MD, Principal Investigator — Tokyo Metropolitan Komagome Hospital
Locations (1):
- Tokyo Metropolitan Komagome Hospital, Bunkyo-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kimura K, Tanuma J, Kimura M, Imamura J, Yanase M, Ieiri I, Kurosaki M, Watanabe T, Endo T, Yotsuyanagi H, Gatanaga H. Safety and tolerability of OP-724 in patients with haemophilia and liver cirrhosis due to HIV/HCV coinfection: an investigator-initiated, open-label, non-randomised, single-centre, phase I study. BMJ Open Gastroenterol. 2024 Apr 27;11(1):e001341. doi: 10.1136/bmjgast-2023-001341. PMID 38677720